CLINICAL TRIAL: NCT02879149
Title: A Prospective, Controlled, Multi-Center, Post-Approval Trial to Evaluate the Long-term Safety and Effectiveness of AUGMENT® Bone Graft Compared to Autologous Bone Graft as a Bone Regeneration Device in Foot and Ankle Fusions
Brief Title: Long-term Safety and Effectiveness of AUGMENT® Bone Graft Compared to Autologous Bone Graft
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BMTI-2015-01
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Ankle and Hindfoot Arthrodesis
Keywords: Ankle Fusions; AUGMENT® Bone Graft; Autologous Bone Graft; arthritis; ankle pain; foot pain; hindfoot fracture; ankle fracture
MeSH Terms: conditions — Arthritis; Ankle Fractures | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples for antibody testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Standard Rigid Fixation plus autograft
  Interventions: Procedure: Standard of Care
- Group 2: Standard rigid fixation plus AUGMENT® Bone Graft
  Interventions: Device: AUGMENT® Bone Graft

INTERVENTIONS:
Device: AUGMENT® Bone Graft — AUGMENT® Bone Graft
  Groups: Group 2
Procedure: Standard of Care — Autologous Bone Graft
  Groups: Group 1

SUMMARY:
The objective of this long-term study is to evaluate the long term effectiveness and safety of AUGMENT® Bone Graft vs. autologous bone graft. The study involves evaluation of subjects originally treated under Protocol BMTI-2006-01.

Subjects will be asked to consent and return to provide long-term follow-up data at or after 60 months (5 years) have elapsed since their original surgery as a subject in protocol BMTI-2006-01.

STUDY HYPOTHESIS: The effectiveness and safety profile for AUGMENT® Bone Graft is maintained and remains comparable to that of autologous bone graft over long-term subject follow-up.

REGULATORY PHASE: Post-approval study

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria may be included in the study:

1. Must be willing and able to provide informed consent and be available for the planned follow-up evaluations and radiologic tests; and
2. Must have been randomized, treated and included in the safety population of Protocol BMTI-2006-01 (see Exhibit 13.1).

Exclusion Criteria:

1) Subjects that were excluded from the safety analysis in the BMTI-2006-01 study (subjects not listed in Exhibit 13.1). These subjects were consented, but never treated as part of the BMTI-2006-01 protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects over the age of 18 years of age, who were randomized and treated as part of the population of the BMTI-2006-01 protocol.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Demonstration of bridging bone via CT | Months 60 or greater
Subject function as determined by pain on weight bearing | Months 60 or greater
Subject function as determined by AOFAS - AHS score | Months 60 or greater
Subject function as determined by Foot Function Index | Months 60 or greater

CONTACTS AND LOCATIONS:
Locations (26):
- United States (21):
  - Tucson Orthopedic Institute, Tucson, Arizona
  - OrthoNorcal, Capitola, California
  - California Pacific Medical Center, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Center for Bone and Joint Surgery, Royal Palm Beach, Florida
  - Illinois Bone and Joint Institute, LLC, Glenview, Illinois
  - MedStar Health Research Institute/ Union Memorial Hospital, Baltimore, Maryland
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - Michigan Orthopedic Center, Lansing, Michigan
  - Desert Orthopaedics, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - OrthoCarolina, Charlotte, North Carolina
  - Duke University Medical, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Orthopedic Foot and Ankle Center / OhioHealth Research Institute, Westerville, Ohio
  - The Center, Bend, Oregon
  - Rothman Institute, Philadelphia, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The Orthopaedic Foot & Ankle Center, Falls Church, Virginia
- Canada (5):
  - Office of Orthopaedic Surgeons, Talisman Centre North Building, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - QEll Health Sciences Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.aofas.org